CLINICAL TRIAL: NCT04902014
Title: The Combined Effect OF Motivational Interviewing and Wearable Fitness Trackers on Motivation and Physical Activity In Inactive Adults: A Randomized Controlled Trial
Brief Title: A Study to Test the Effectiveness of Different Interventions to Improve Physical Activity in Adults.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 19-9439H
Record Dates: First submitted 2021-05-09; First posted 2021-05-26 (Actual); Results first posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2022-09

CONDITIONS: Healthy
Keywords: mHealth; physical activity; motivation; self-determination theory
MeSH Terms: conditions — Motor Activity | interventions — Motivational Interviewing; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Education (Active Comparator)
  Interventions: Behavioral: Education
- Motivational Interviewing (Experimental)
  Interventions: Behavioral: Motivational Interviewing
- Wearable Fitness Tracker (Experimental)
  Interventions: Behavioral: Wearable Fitness Trackers
- Wearable Fitness Tracker+ (Experimental)
  Interventions: Behavioral: Wearable Fitness Tracker+

INTERVENTIONS:
Behavioral: Motivational Interviewing — The individuals will be scheduled for and participate in six biweekly in person SDT based MI sessions. These sessions will take place in the HPCRL at CSU. The MI sessions will be conducted by a PhD student who has been trained by a MI practitioner. Participants will be provided a log book and will be asked to log their PA, with the goal of completing at least 150 minutes of PA per week. They will set biweekly PA goals, which will be discussed in the MI sessions. These participants will also receive general physical activity guidelines education and information on strategies to reach the recommended amount of activity per week during the initial baseline assessment meeting.
  Arms: Motivational Interviewing
Behavioral: Education — These participants will receive general physical activity guidelines education and information on strategies to reach the recommended amount of activity per week during the initial baseline assessment meeting. These participants will not do any other study related activities. At the conclusion of the study, these participants will be offered the chance to participate in one MI session.
  Arms: Education
Behavioral: Wearable Fitness Trackers — Individuals assigned to this experimental condition will be given a wrist-worn WFT and will be instructed to wear it for the duration of the study. They will also download the corresponding mobile application on their smartphones. They will be trained by a member of our team on how to utilize the WFT and mobile application. The intended WFT tracks daily steps, miles traveled, kcals expended, and daily activity time. This device provides these data to the wearer via a small screen. Participants will be instructed to aim to complete at least 150 minutes of PA per week. Researchers will have the capability to track participant daily PA via the WFT and associated API. These individuals will be asked to set biweekly PA goals. These participants will also receive general physical activity guidelines education and information on strategies to reach the recommended amount of activity per week during the initial baseline assessment meeting.
  Arms: Wearable Fitness Tracker
Behavioral: Wearable Fitness Tracker+ — These individuals will be given the wrist-worn WFT, be instructed to wear it for the duration of the study AND be scheduled for six SDT based MI sessions. These participants will also be trained by a member of our team on how to utilize the WFT and associated application. They will be instructed to aim to complete 150 minutes of PA per week. These participants will be asked to set biweekly PA goals which will be discussed in MI sessions. Researchers will have the capability to track participant daily PA via the WFT and associated API. These participants will also receive general physical activity guidelines education and information on strategies to reach the recommended amount of activity per week during the initial baseline assessment meeting.
  Arms: Wearable Fitness Tracker+

SUMMARY:
During the initial months of the COVID-19 pandemic, physical activity (PA) engagement levels declined worldwide. Despite the overwhelming adoption of wearable fitness tracker (WFT) devices, it continues to be unclear as to their effect on PA engagement or PA motivation. Building on past research, we hypothesized that combining a WFT with a known impactful intervention, motivational interviewing (MI) would positively influence both self-determination theory (SDT) motivation and PA during an unprecedented global emergency.

A four-group randomized controlled study was conducted amongst 40 inactive adults over a 12-week period during the COVID-19 pandemic. One group (WFT, n = 10) received a wearable fitness tracker, a second (MI, n=10) received bi-weekly MI sessions, a third (WFT+, n=10) received both, and a fourth (Education, n=10) received basic PA education. Outcome measures for motivation and PA were measured though an online survey before and after the 12-week period.

ELIGIBILITY:
Inclusion Criteria:

* Females or males, aged 18 or older,
* does not currently engage in 150 minutes of moderate to vigorous PA per week,
* owns an Android, or iPhone smartphone device,
* is willing to download a mobile app to be used on the smartphone device, 5) is willing to wear a small, wrist worn fitness tracker for the duration of the study, and 6) is be willing to attend 6 biweekly MI sessions over 12 weeks.

Exclusion Criteria:

* a history of myocardial infarction, angina, coronary artery bypass surgery, congestive heart failure, or diabetes,
* limiting conditions such as concurrent cancer treatment, peripheral artery disease, orthopedic injury, or pain limiting arthritis,
* seeking to participate in other structured PA programs during the duration of the study,
* pregnant at the initiation of the study or plans to become pregnant during the study, and
* alcohol or other substance abuse within the previous 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-04-13 (Actual); Primary Completion 2020-09-21 (Actual); Study Completion 2020-09-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Human Performance Clinical Research Laboratory, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through a variety of means including flyers on the Colorado State University campus, social media, and mass emails. Participants were recruited and admitted into the study on a rolling basis from April 2020-June 2020.
Pre-assignment Details: Consented participants were stratified by sex (male/female) and age (20-29, 30-39, 40-49, 50-59, and 60-69 y/o.) before being randomized to one of four conditions.
Period: Overall Study
Arm/Group | Education | Motivational Interviewing | Wearable Fitness Tracker | Wearable Fitness Tracker+
Started | 10 | 10 | 10 | 10
Completed | 10 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Education | Motivational Interviewing | Wearable Fitness Tracker | Wearable Fitness Tracker+ | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 10 | 10 | 40
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.8 (12.80) | 40.0 (11.27) | 42.3 (12.21) | 42.4 (10.08) | 41.6 (11.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 8 | 8 | 32
  Male | 2 | 2 | 2 | 2 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 8 | 10 | 10 | 8 | 36
  Unknown or Not Reported | 2 | 0 | 0 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 10 | 9 | 10 | 10 | 39
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 10 | 40
Income [Count of Participants; unit: Participants]
  $12,500-$26,999 | 0 | 0 | 1 | 0 | 1
  $27,000-$43,999 | 1 | 2 | 1 | 0 | 4
  $44,000-$59,999 | 1 | 0 | 1 | 4 | 6
  $60,000-$74,999 | 2 | 1 | 2 | 1 | 6
  $75,000-$99,999 | 2 | 1 | 1 | 0 | 4
  $100,000-$150,000 | 2 | 5 | 1 | 3 | 11
  More than $150,000 | 2 | 1 | 2 | 1 | 6
  Do Not Know/Prefer Not to Answer | 0 | 0 | 1 | 1 | 2
Education [Count of Participants; unit: Participants]
  High School or GED | 0 | 0 | 0 | 1 | 1
  Some College | 0 | 2 | 0 | 0 | 2
  College Degree | 5 | 1 | 3 | 2 | 11
  Graduate Degree | 5 | 7 | 7 | 7 | 26
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 28.89 (6.81) | 28.31 (5.01) | 25.68 (4.54) | 30.53 (7.23) | 28.35 (5.90)
Motivation Variables [Mean (Standard Deviation); unit: units on a scale] — The Behavioral Regulations in Exercise Scale version 3, (BREQ-3) was used to collect pre- and post- motivation for exercise variables including Amotivation, External, Introjected, Identified, and Integrated Regulation, and Intrinsic Motivation. The scale is on a 0 (does not apply to me) to 4 (applies to me very much) scale.
  The Basic Psychological Needs in Exercise Scale was used to collect pre- and post- autonomy, competence, and relatedness. The scale is on a 0 (does not apply to me) to 4 (applies to me very much) scale.
  units on a scale
    Amotivation | 0.48 (0.48) | 0.48 (0.46) | 0.35 (0.41) | 0.83 (0.31) | 0.54 (0.42)
    External Regulation | 1.43 (1.06) | 1.83 (1.04) | 0.98 (0.32) | 1.53 (0.78) | 1.44 (0.80)
    Introjected Regulation | 2.17 (0.82) | 2.35 (1.07) | 2.23 (0.95) | 2.62 (0.63) | 2.34 (0.87)
    Identified Regulation | 3.06 (0.65) | 2.60 (0.49) | 3.10 (0.52) | 2.98 (0.32) | 2.94 (0.50)
    Integrated Regulation | 2.09 (0.57) | 1.73 (0.51) | 2.50 (0.94) | 2.03 (0.49) | 2.09 (0.61)
    Intrinsic Regulation | 2.07 (0.73) | 1.98 (0.82) | 2.53 (1.07) | 1.83 (0.89) | 2.10 (0.88)
    Relative Autonomy Index | 3.13 (2.78) | 1.65 (2.06) | 4.57 (3.03) | 4.78 (2.22) | 3.53 (2.52)
    Autonomy | 3.60 (0.35) | 3.28 (0.52) | 3.68 (0.56) | 3.63 (0.51) | 3.55 (0.49)
    Competence | 3.10 (0.64) | 2.78 (0.48) | 3.03 (1.22) | 2.62 (0.73) | 2.88 (0.77)
    Relatedness | 3.08 (0.58) | 3.35 (0.76) | 3.00 (0.37) | 3.30 (0.86) | 3.18 (0.63)
Physical Activity Variables [Mean (Standard Deviation); unit: units on a scale]
  Minutes of Moderate to Vigorous Physical Activity per Day | 65.37 (19.82) | 56.26 (25.10) | 74.05 (23.58) | 53.82 (20.88) | 62.38 (22.35)
  Minutes of Moderate to Vigorous Physical Activity Minutes per Weekday | 62.55 (22.43) | 51.63 (26.84) | 74.18 (32.55) | 51.90 (22.18) | 60.07 (26.08)
  Minutes of Moderate to Vigorous Physical Activity Minutes per Weekend Day | 73.25 (30.61) | 69.16 (38.20) | 70.58 (18.33) | 63.87 (27.17) | 69.22 (28.71)
  Steps per Day | 5690.71 (1974.24) | 4640.30 (1759.94) | 5817.82 (2334.36) | 5564.56 (1783.55) | 5428.35 (1963.02)
  Steps per Weekday | 5322.45 (2101.10) | 4514.95 (2646.50) | 5877.11 (2741.19) | 5346.10 (1712.86) | 5265.15 (2300.41)
  Steps per Weekend Day | 6449.33 (3056.45) | 5293.85 (2554.78) | 5494.35 (2142.58) | 6189.68 (2784.17) | 5856.80 (2634.49)

OUTCOME MEASURES:

1. Primary Outcome: Change in Motivation From Baseline at 12 Weeks.
Description: Changes in motivation for physical activity as described by the self-determination theory was assessed using the Behavioral Regulation in Exercise Questionnaire, v3 (BREQ-3) and the Basic Psychological Needs in Exercise Scale (BPNS). The BREQ-3 uses four survey items per motivational subtype (Amotivation, External, Introjected, Identified, and Integrated Regulation, and Intrinsic Motivation). The BPNS uses three of four items per psychological need (Autonomy, Competence, and Relatedness) The raw scores per subtype or need are averaged for one subtype and need score per participant. The scale ranges from 0 (does not apply to me) to 4 (applies to me very much). Therefore, subtype or need score closer to ) indicate low levels of that subtype whereas scores closer to 4 indicate higher levels of that subtype or need.
Time Frame: Baseline and at 12 weeks.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Education | Motivational Interviewing | Wearable Fitness Tracker | Wearable Fitness Tracker+
Number analyzed (Participants) | 10 | 10 | 10 | 10
Units on a scale
  Amotivation | 0.30 (0.40) | 0.48 (0.43) | 0.40 (0.36) | 0.43 (0.49)
  External Regulation | 1.58 (1.25) | 1.45 (0.91) | 0.89 (0.40) | 1.27 (0.73)
  Introjected Regulation | 2.45 (1.02) | 2.33 (0.82) | 2.31 (0.77) | 2.48 (0.63)
  Identified Regulation | 3.10 (0.47) | 3.10 (0.53) | 3.20 (0.75) | 3.33 (0.54)
  Integrated Regulation | 2.38 (0.93) | 2.45 (0.47) | 2.61 (0.81) | 2.63 (0.83)
  Intrinsic Motivation | 2.47 (0.53) | 2.70 (0.62) | 2.87 (0.80) | 2.98 (0.59)
  Relative Autonomy Index | 3.37 (2.59) | 4.00 (2.06) | 5.08 (2.27) | 4.78 (2.22)
  Autonomy | 3.62 (0.72) | 3.97 (0.43) | 4.10 (0.45) | 4.23 (0.35)
  Competence | 3.20 (0.83) | 3.83 (0.33) | 3.65 (0.97) | 3.75 (0.68)
  Relatedness | 3.06 (1.18) | 3.92 (0.68) | 3.14 (0.26) | 3.87 (0.67)

2. Primary Outcome: Change in Moderate to Vigorous Physical Activity From Baseline at 12 Weeks.
Description: Moderate to Vigorous Physical Activity (MVPA) was assessed using five days (4 weekdays and 1 weekend day) of actigraphy (ActiGraph).
Time Frame: Baseline and at 12 weeks
Measure: Mean (Standard Deviation); unit: Minutes of MVPA per day
Arm/Group | Education | Motivational Interviewing | Wearable Fitness Tracker | Wearable Fitness Tracker+
Number analyzed (Participants) | 10 | 10 | 10 | 10
Minutes of MVPA per day
  Minutes of Moderate to Vigorous Physical Activity per Day | 66.70 (17.83) | 67.75 (16.47) | 76.37 (29.19) | 71.08 (36.90)
  Minutes of Moderate to Vigorous Physical Activity per Weekday | 66.17 (16.99) | 64.00 (25.10) | 78.97 (32.67) | 68.60 (41.11)
  Minutes of Moderate to Vigorous Activity per Weekend Day | 72.32 (29.27) | 69.70 (22.30) | 66.17 (38.62) | 76.38 (38.50)

3. Primary Outcome: Change in Steps Per Day From Baseline at 12 Weeks.
Description: Steps per day was assessed using five days (4 weekdays and 1 weekend day) of actigraphy (ActiGraph).
Time Frame: Baseline and at 12 weeks
Measure: Mean (Standard Deviation); unit: Steps per day
Arm/Group | Education | Motivational Interviewing | Wearable Fitness Tracker | Wearable Fitness Tracker+
Number analyzed (Participants) | 10 | 10 | 10 | 10
Steps per day
  Steps per Day | 6155.58 (1370.35) | 5400.56 (1314.90) | 6693.01 (2394.24) | 6232.15 (2857.27)
  Steps per Weekday | 6216.31 (1370.35) | 5211.16 (1847.80) | 7183.81 (2430.83) | 6123.24 (3047.30)
  Steps per Weekend Day | 6387.75 (2350.78) | 5235.22 (1749.21) | 5275.90 (3292.88) | 6565.06 (3156.44)

ADVERSE EVENTS:
Time Frame: Twelve weeks
Arm/Group | Education | Motivational Interviewing | Wearable Fitness Tracker | Wearable Fitness Tracker+
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
Conducted the study during the COVID-19 pandemic. Homogenous sample. Did not assess wear time or compliance with wear directives in WFT and WFT+ groups. RAI does not allow for an investigation into the more nuanced and multidimensional aspects of SDT motivation as it pertains to PA.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-08): https://cdn.clinicaltrials.gov/large-docs/14/NCT04902014/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-08): https://cdn.clinicaltrials.gov/large-docs/14/NCT04902014/ICF_001.pdf